CLINICAL TRIAL: NCT01171092
Title: A Pilot Trial to Assess Mobilization of Hematopoietic Progenitor Cells With a Combination of Bortezomib and G-CSF in Patients Undergoing Autologous Transplant for Myeloma and Lymphoma
Brief Title: A Safety Study Looking at the Combination of Velcade and G-CSF in Patients With Myeloma or Lymphoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11803; X05279 (Other: Millenium Pharmaceuticals)
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Malignant Lymphoma, Stem Cell Type; Autologous Transplant
Keywords: stem cell; transplant; myeloma; lymphoma; BMT; autologous
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell | interventions — Bortezomib; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib and G-CSF (Experimental)
  Interventions: Drug: bortezomib and G-CSF

INTERVENTIONS:
Drug: bortezomib and G-CSF — Bortezomib injection:
  1.3mg/m2 11 days before and 8 days before the stem cell collection
  G-CSF injection:
  10mcg/kg on days -4 to day -1 once daily
  Other Names: Velcade; Filgrastim

SUMMARY:
The purpose of this study is to determine if the combination of G-CSF and bortezomib is safe and effective in blood cell mobilization.

DETAILED DESCRIPTION:
The study plans to use VELCADE for two doses followed by G-CSF given for 4 doses as is standard for mobilization with G-CSF alone. The rationale for VELCADE prior to the G-CSF is because VELCADE causes thrombocytopenia, similar to how cyclophosphamide is given followed by G-CSF for stem cell mobilization. Usually a cycle of VELCADE for myeloma therapy consists of 4 doses, but this may result in more significant drop in the platelet count. Low platelet counts may preclude adequate stem cell collection. The mobilization with VELCADE and GCSF will be approximately 3 -4 weeks after completion of the initial therapy for the primary disease.

Patients meeting eligibility criteria and who give informed consent will be mobilized using bortezomib at 1.3mg/m2 on day -11 and day -8. Subsequently G-CSF will be administered subcutaneously from day -4 to day -1 as a once daily injection at the standard /established dose of 10mcg/kg. Stem cell collection will be done on day 0 per standard of care regimen and protocol with processing of 4 -5 blood volumes. Stem cell enumeration by flow cytometry will be done prior to the collection by flow cytometry. The number of CD 34 positive cells (stem cell phenotype) / kg obtained each day of collection will be noted. G-CSF will be continued daily until adequate numbers of stem cells are obtained for the performance of a single autologous transplant (> 2.5 million CD 34 cells/kg of weight. Subsequently the data for engraftment of neutrophils and platelets will be monitored as is routine for all patients undergoing autologous transplant.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal for at least 1 year before the screening visit, or surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse.
* Male subject, even if surgically sterilized (ie, status post vasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* > 18 yrs of age needing to undergo an autologous blood stem cell transplant for the treatment of multiple myeloma or lymphoma

Exclusion Criteria Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patient has a platelet count of < 100x 109/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of < 1.0x109/ within 14 days before enrollment.
* Patient has > 1.5 x ULN Total Bilirubin
* Patient has a calculated or measured creatinine clearance of < 50 mL/minute within 14 days before enrollment.
* Patient has ≥ Grade 2 peripheral neuropathy.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to VELCADE, boron or mannitol or G-CSF
* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial until 2 weeks after patient has received the last dose of Velcade for mobilization.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Treated with VELCADE in the past 30 days
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness of the combination of bortezomib and G-CSF | 100 days after transplant
  The primary aim of this single-arm pilot study is to determine the effectiveness of a combination of Bortezomib and G-SCSF in blood stem cell mobilization through the estimation of the proportion of patients receiving treatment that obtain adequate stem cell yield.

SECONDARY OUTCOMES:
Assess the safety of the combination of bortezomib and G-CSF | 365 days after transplant
  Assess the safety of the study mobilization regimen

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Abhyankar, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Westwood Campus, Westwood, Kansas